CLINICAL TRIAL: NCT00136578
Title: A Phase I, Open-Label, Dose-Escalation Study of the Safety and Tolerability of Ispinesib in Combination With Carboplatin on an Every 21-Day Schedule in Subjects With Advanced Solid Tumors.
Brief Title: Ispinesib In Combination With Carboplatin In Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSP10014
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Solid Tumours
Keywords: solid tumors; dose limiting toxicity; carboplatin; tolerability; Safety
MeSH Terms: interventions — ispinesib; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subjects receiving carboplatin and SB-715992 (Experimental): Subjects will receive carboplatin on Day 1 as an intravenous (IV) infusion over 30 minutes followed by 1-hour IV infusion of SB-715992 once every 21 days.
  Interventions: Drug: SB-715992; Drug: carboplatin

INTERVENTIONS:
Drug: SB-715992 — SB-715992 will be available either as 5 milliliter (mL) vial containing 4 milligram (mg) of SB-715992 or 4 mL vial containing 5 mg of SB-715992 at a concentration of 1 mg/mL OR a 10 mL vial that contains 10 mg of SB-715992 in a 10 mL solution at a concentration of 1 mg/mL.
Drug: carboplatin — Carboplatin will be available as sterile, lyophilized white powder available in single-dose vials containing 50 mg, 150 mg, and 450 mg of carboplatin for administration by IV infusion. Each vial will be reconstituted with either Sterile Water for Injection, USP, 5% Dextrose in Water (D 5 W), or 0.9% Sodium Chloride Injection, USP.

SUMMARY:
The purpose of this study is to determine the dose regimen of Ispinesib in combination with carboplatin in patients with solid tumors. Ispinesib is dosed by 1-hour intravenous infusion and carboplatin is dosed by 30 minute intravenous infusion every 3 weeks (on the same day). A patient may continue to receive treatment as long as they are benefiting from the treatment. Blood samples will be taken at specific times to measure the amount of both drugs in your body at specific times after the drug is given. Blood samples will also be taken for lab tests such as complete blood counts and clinical chemistries. Physical exams will be performed before each treatment with Ispinesib. During the treatment phase, the patients will undergo regular assessments for safety and clinical response.

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically confirmed diagnosis of an advanced solid tumor malignancy that is not responsive to standard therapies or for which there is no standard therapy.
* ECOG (Eastern Cooperative Oncology Group) Performance Status of 0-2.

Exclusion criteria:

* Females who are pregnant or nursing.
* Pre-existing hemolytic anemia.
* Pre-existing peripheral neuropathy greater than or equal grade 2. Greater than or equal to 4 prior chemotherapy regimens including neoadjuvant/adjuvant chemotherapy, except breast cancer subjects who may have received more than 4 prior chemotherapy regimens.
* Absolute neutrophil count less than 1,500/mm3.
* Platelets less than 100,000/mm3.
* Hemoglobin less than 9 g/dL.
* Total bilirubin greater than1.5 mg/dL.
* AST/ALT greater than 2.5 X upper limit of normal.
* Creatinine clearance less than or equal to 50 mL/min (calculated by the Cockcroft Gault Formula).
* Known contra-indications to the use of carboplatin, cisplatin, or other platinum-containing compounds.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-10-20 (Actual); Primary Completion 2006-10-25 (Actual); Study Completion 2006-10-25 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability endpoints will consist of the valuation of adverse events (AEs),vital signs and laboratory values. A dose regimen where = 1 of 6 (or =17%) subjects experience a dose-limiting toxicity. | Up to Day 154

SECONDARY OUTCOMES:
Antitumor activity will be assessed every 2 cycles and will be recorded as complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD). | Up to 140

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Nashville, Tennessee, United States
- GSK Investigational Site, Newcastle upon Tyne, Northumberland, United Kingdom

REFERENCES:
- See also: Results for study KSP10014 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/KSP10014?search=study&search_terms=KSP10014#rs